CLINICAL TRIAL: NCT00462046
Title: The Efficacy and Safety of Berberine in the Treatment of Type 2 Diabetes With Dyslipidemia
Brief Title: Efficacy and Safety of Berberine in the Treatment of Diabetes With Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CCEMD001
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus, Type 2; Metabolic Syndrome
Keywords: Berberine; Type 2 diabetes; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Dyslipidemias | interventions — Berberine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Berberine

SUMMARY:
Berberine has showed effective in lowering blood sugar levels in db/db mice and anti-dyslipidemia in human. These findings have not been tested in a clinical trial. This randomized, double blind, placebo controlled and multi-center study has demonstrated that berberine is effective in lowering plasma glucose concentrations, reducing serum HbA1c and anti-dyslipidemia in type 2 diabetic patients with dyslipidemia.

DETAILED DESCRIPTION:
Berberine, a natural plant alkaloid, has not been well investigated for clinical application in the treatment of diabetes. The present study evaluated the efficacy and safety of berberine in the treatment of type 2 diabetic patients with dyslipidemia. 116 patients with type 2 diabetes and dyslipidemia were assigned in a randomized, double-blind, and placebo-controlled 4-clinical center study to receive berberine (1.0g daily) or placebo for 3 months. The primary efficacy outcomes were changes in plasma glucose and serum lipid levels. The glucose disposal rate (GDR) was measured using a hyperinsulinemic euglycemic clamp to assess insulin resistance in a randomly selected subjects of 54 patients. The baseline characteristics were similar in berberine and placebo groups. After 3 months, fasting and post load plasma glucose levels, HbA1C, triglyceride, total cholesterol and LDL-C levels were all significantly reduced in the berberine group compared with the placebo group (p<0.0001, p<0.0001, p<0.0001, p=0.002, p<0.0001 and p<0.0001 respectively). The GDR was significantly increased after 3 months of berberine (p=0.037), while no change was found in the placebo group (p=0.86). BMI, systolic blood pressure and serum IL-6 levels were all significantly reduced after treatment in berberine group as compared with the placebo group (p=0.016, p=0.041 and p=0.014, respectively). Our results show berberine to be effective and safe in the treatment of persons with diabetes and dislipidemia. This agent may be useful in the treatment of patients with type 2 diabetes, and could play a role in treatment of metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 25 -70 years;
2. Newly diagnosed type 2 diabetes according to the 1999 World Health Organization criteria;
3. Dyslipidemia with TG> 150mg/dL (1.70mmol/L), and/or TC>200mg/dL (5.16mmol/L), and/or LDL-C>100mg/dL (2.58mmol/L) according to the National Cholesterol Education Program's Adult Treatment Panel III (NCEP: ATPIII) without previous treatment.
4. BMI:19 - 40 kg/m2.

Exclusion Criteria:

1. Moderate or severe liver or renal dysfunction, psychiatric disease or severe infection;
2. Severe dysfunction of the heart，New York Heart Association class ³ Ⅲ phase;
3. History of acute diabetic complications;
4. Pregnancy or planned pregnancy.
5. Present or previous use of drugs for treatment of diabetes or dyslipidemia;
6. Fasting plasma glucose >8mmol/L and/or post load plasma glucose level >17mmol/L after 2-week run-in.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-04; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Fasting glucose levels
OGTT 2h glucose levels
HbA1c
Serum Triglycerides
Serum Total Cholesterol
HDL-c
LDL-c

SECONDARY OUTCOMES:
Glucose Disposal Rate
BMI
Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Ying Li, MD,PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine